Official Title: Assessing patient confidence in biologic medications (research study vs anecdotal

evidence) NCT03168347

IRB Approval Date: 05/11/2018

# **Assessing Patient Confidence in Biologic Medication**

Study Fact Sheet

Steven R. Feldman, M.D., Ph.D., Principal Investigator

#### Introduction

You are receiving this document because you have been/will be seen by a dermatologist at Wake Forest Baptist Hospital. We would like to invite you to participate in a research study that will help us better understand the experiences of patients with psoriasis in our community.

#### Why Is This Study Being Done?

The purpose of this research study is to learn more about patient's perception of certain psoriasis treatment options.

## How Many People Will Take Part in the Study?

400 people at 1 research site will take part in this study.

## What Is Involved in the Study?

We would like for you to answer a few questions about your willingness to use psoriasis medication. This survey includes up to eight questions and will take approximately one minute to complete. The survey is anonymous; no identifying information will be collected.

#### How Long Will I Be in the Study?

You will be in the study for 1 day.

## What Are My Rights as a Research Study Participant?

It is important that you know that this document is not to tell you to join this study. It is your decision. Your participation is voluntary. While we hope you will consider participating, whether or not you participate in this study will have no effect on your relationship with Wake Forest Baptist Health as a patient.

# WHOM DO I CALL IF IHAVE QUESTIONS OR PROBLEMS?

| This is an approved Institutional Review Board (IRB) research study: # IRB00043948. For questions about the |
|---|
| study contact the study investigator, Steven R. Feldman, M.D., Ph.D. at |
| or The Institutional Review Board (IRB) a group of people who review the |
| research to protect your rights. If you have a question about your rights as a research participant, or you would |
| like to discuss problems or concerns, have questions or want to offer input, or you want to obtain additional |
| information, you should contact the Chairman of the IRB at .Completion of the survey implies |
| your consent to participate in the study. With your participation in this survey, you can help us learn more about |
| psoriasis! We thank you kindly for your time. If you have any further questions about this survey, please do not |
| hesitate to contact our study coordinator Irma Richardson at or Email: |